CLINICAL TRIAL: NCT04717388
Title: Cognitive and Emotional Function and Brain Reorganisation Associated to Auditory Abilities : Impact of Tinnitus
Brief Title: Pathophysiology, Psycho-emotional and Cognitive Functioning Associated With Tinnitus
Acronym: AudiCog
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP200761
Record Dates: First submitted 2020-12-15; First posted 2021-01-22 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Tinnitus; Epilepsy, Temporal Lobe
Keywords: Tinnitus; Epilepsy; Cognitive Functioning; Brain connectivity
MeSH Terms: conditions — Tinnitus; Epilepsy, Temporal Lobe; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- impact of tinnitus on executive cognitive functioning (Experimental)
  Interventions: Other: acoustics tests, Questionaries,
- impact of tinnitus on reorganization of functional/ structural brain connectivity maps (Experimental)
  Interventions: Other: acoustics tests, Questionaries,; Radiation: MRI

INTERVENTIONS:
Other: acoustics tests, Questionaries, — acoustics tests at V1 Questionaries at V1
  * cognitive
  * emotional
  * auditory
Radiation: MRI — Anatomical and functional MRI at V2
  Arms: impact of tinnitus on reorganization of functional/ structural brain connectivity maps

SUMMARY:
the investigators have recently shown that patients with drug-resistant temporal lobe epilepsy who have undergone brain surgery targeting the medial temporal lobe structures were more likely to develop tinnitus postoperatively. This discovery of a vulnerability to tinnitus associated with medial temporal lobe surgery to eliminate drug-refractory epileptic seizures provides a new clinical model of tinnitus, targeting temporal lobe regions as generators or mediators of this hearing disorder. The objective of this project is to study the impact of tinnitus on the cognitive, emotional, psychoacoustic and cerebral functioning associated with this hearing disorder, and to clarify the pathophysiology of tinnitus by comparing different groups of individuals with tinnitus (surgical epileptic patients or non-surgical ORL patients) to matched tinnitus-free groups (surgical tinnitus-free cases and healthy controls volunteer).

DETAILED DESCRIPTION:
Tinnitus (known as "ringing in the ears") is a disabling medical condition. Its psychosocial impact is substantial, including anxiety, depression, stress, irritability, concentration and sleep disorder leading to detrimental effects on communication, education, professional fulfillment, mental health and quality of life. The cerebral bases of tinnitus and its consequence on human hearing health have received a lot of attention in the scientific literature. Yet, the relationship between the neurobiological dysfunction, psychological processes and clinical semiology of tinnitus remains poorly understood. Considering the current gaps in knowledge, there is a real need for clinical investigations into tinnitus-related brain changes and rigorous hearing, psycho-emotional, and cognitive assessments. the investigators recent discovery of a vulnerability to tinnitus associated with medial temporal lobe surgery (to treat refractory epilepsy) provides a new clinical model, which targets the temporal lobe regions as a tinnitus generator or mediator of its severity. The goal of this collaborative interdisciplinary study is to advance knowledge about the pathophysiology of tinnitus, as well as the socio-emotional, cognitive and psychoacoustic aspects associated to this hearing disorder. the investigators will first, characterize the subjective and self-reported hearing disorders with objective psychoacoustic, cognitive and affective measures in tinnitus sufferers and second, clarify the cerebral network underlying tinnitus and elucidate the role temporal lobe regions in the brain networks at play in surgical and non-surgical tinnitus. To this end, individuals with and without tinnitus, who had undergone or not a surgery will be compared in a 2 by 2 design. Investigating different patient cohorts with tinnitus who are well matched to both, healthy control populations and vulnerable clinical populations, without tinnitus is a valuable contribution of our proposal. Moreover, the psychological and hearing profiles of people with tinnitus will be examined in relation with their brain morphology and connectivity profiles.The project builds upon the internationally recognized leadership of the PI and her collaborators in the fields of auditory cognition and its neurobiological bases using neuropsychological, psychoacoustic, and neuroimaging methods in clinical populations. The members of the investigators consortium have all the necessary and unique expertise to carry out this innovative and interdisciplinary project.

ELIGIBILITY:
Common Criteria for Inclusion :

* Age ≥ 18 years old
* Good written and oral comprehension of the French language
* Person affiliated to a Social Security scheme
* Informed consent signed by the participant
* Normal or corrected vision
* Absence of known pre-existing neurological and/or degenerative disorders

Group Specific Inclusion Criteria :

Tinnitus+ Group - Suffering from subjective uni- or bilateral tinnitus, chronic (>3 months) and stable (no period of remission).

Chir+ Group

- Surgically treated for drug-resistant epilepsy of the temporal lobe (including the amygdala).

Group Tinnitus-

* Not suffering from tinnitus Group Chir-
* Non epileptic
* Not having undergone surgical treatment of the temporal lobe (including the tonsil)

Exclusion criteria:

* Presence of severe or profound deafness, uni or bilateral.
* Under legal protection (guardianship, curators, etc.)

Additional criteria for patients completing visit V2 :

* MRI contraindicated or claustrophobic
* Pregnant or breastfeeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2027-10-15 (Estimated); Study Completion 2029-04-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the impact of tinnitus on executive cognitive functioning | at the second visit, maximum 6 month after first visit.
  Measurement of executive control using a stroop test in people with and without chronic tinnitus.

SECONDARY OUTCOMES:
Emotional functioning (anxiety and depression) | at the second visit, maximum 6 month after first visit.
  Measures of Anxiety and Depression using: Hospital Anxiety and Depression Scale (HADS) : 14 rated items from 0 to 3. Seven questions are related to anxiety and seven to the depressive dimension, allowing for thus obtaining two scores (maximum score of each score = 21).
psycho-acoustic functioning | at the second visit, maximum 6 month after first visit.
  Measurements of auditory functioning through hearing assessment (audiometry) :
  - Self-assessment questionnaires for hearing loss: The self-assessment of hearing loss is based on a yes/no question: "Do you feel that you have a hearing loss or hearing loss?
psycho-acoustic functioning | at the second visit, maximum 6 month after first visit.
  Measurements of auditory functioning through hearing assessment (audiometry) :
  - The noise hypersensitivity questionnaire( Khalfa, 2002) provides a score ranging from 0 (no hypersensitivity) to 42 (very strong hypersensitivity).
psycho-acoustic functioning | at the second visit, maximum 6 month after first visit.
  Measurements of auditory functioning through hearing assessment (audiometry) :
  - The severity of tinnitus is measured by the Tinnitus Handicap Inventory (THI) questionnaire. Scores range from 0 (mild discomfort) to 100 (catastrophic impact).
psycho-acoustic functioning | at the second visit, maximum 6 month after first visit.
  Measurements of auditory functioning through hearing assessment (audiometry) :
  - Hearing threshold measurement (pure tones from 125-16000Hz)
psycho-acoustic functioning | at the second visit, maximum 6 month after first visit.
  Measurements of auditory functioning through hearing assessment (audiometry) :
  - Discomfort threshold measurement (with 1kHz sound)
psycho-acoustic functioning | at the second visit, maximum 6 month after first visit.
  Measurements of auditory functioning through hearing assessment (audiometry) : Evaluation of transient otoacoustic emissions (TEOAE) or by distortion product (DPOAE)
cognitive functioning, other than executive functioning (attention, memory) | at the second visit, maximum 6 month after first visit.
  Measures of cognitive functioning :
  - the Attentional Network Test (ANT) visual attention test.
  ANT gives three attention scores based on reaction times. These scores represent the ability to direct attention, to be alert to surrounding stimuli and the executive part of attention.
cognitive functioning, other than executive functioning (attention, memory) | at the second visit, maximum 6 month after first visit.
  Measures of cognitive functioning :
  - Mental Flexibility Score (Trail Making Test): The scores of the TMT (Trail Making Test) are expressed in time of completion. The faster the time to completion, the better the performance. So we have 2 scores, one for board A of the test: TMT-A and the other for board B of the test: TMT-B.
cognitive functioning, other than executive functioning (attention, memory) | at the second visit, maximum 6 month after first visit.
  Measures of cognitive functioning :
  Measures of cognitive functioning :- Short-term memory score (auditive-verbal span). Score between 1 and 10, where 10 represents the best short-term memory score
cognitive functioning, other than executive functioning (attention, memory) | at the second visit, maximum 6 month after first visit.
  Measures of cognitive functioning :
  Measures of cognitive functioning :- Working memory score (Brown-Peterson). The Brown Peterson gives a memorization score ranging from 0 to 100, where 100% is the best score.
cognitive functioning, other than executive functioning (attention, memory) | at the second visit, maximum 6 month after first visit.
  Measures of cognitive functioning :
  - Episodic memory score in auditory modality. The episodic memory test in auditory mode gives a memorization score ranging from 0 to 100, where 100% represents a perfect memorization score.
the reorganization of functional and structural brain connectivity maps | at the third visit, maximum 18 month after the first visit
  Functional and structural brain connectivity measurements using brain imaging (fMRI, diffusion and resting MRI) :
  - Volumetric measurement (in particular of the amygdala and the parahippocampal cortex)
the reorganization of functional and structural brain connectivity maps | at the third visit, maximum 18 month after the first visit
  Functional and structural brain connectivity measurements using brain imaging (fMRI, diffusion and resting MRI) :
  - Measurement of anatomical connections between regions of interest (i.e. amygdala, auditory cortex, attention network including the precuneus and prefrontal cortex) from diffusion tensor imaging (TDI): fractional anisotropy (FA), mean diffusivity (MD), radial (RD) and axial (AD).
the reorganization of functional and structural brain connectivity maps | at the third visit, maximum 18 month after the first visit
  Functional and structural brain connectivity measurements using brain imaging (fMRI, diffusion and resting MRI) :
  - Measurement of structural connectivity from fMRI at rest between predefined regions of interest and over new regions of interest defined during an attentional activation task
the reorganization of functional and structural brain connectivity maps | at the third visit, maximum 18 month after the first visit
  Functional and structural brain connectivity measurements using brain imaging (fMRI, diffusion and resting MRI) :
  - Measurement of the amplitude of the synchrony of slow fluctuations and statistical dependencies in functional connectivity by comparing data from people with and without chronic tinnitus.
Emotional functioning (stress) | at the second visit, maximum 6 month after first visit.
  Measures of stress using Perceived Stress Scale (PSS-4): Lowest score: 0, Highest score: 16, Higher scores are correlated to more stress.
Emotional functioning (Auditory recognition of emotions) | at the second visit, maximum 6 month after first visit.
  Measures of Auditory recognition of emotions using hearing tests with recordings

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Dupont, MD, Ph.D, Study Director — AP-HP Hopital Pitié-Salpêtrière
Locations (2):
- France (2):
  - Service de Soins de Suite et Réadaptation (SSR) Neurologique, DMU de Neurosciences, Paris
  - Hôpital Européen Georges Pompidou, Paris

IPD SHARING:
Plan to Share IPD: No